CLINICAL TRIAL: NCT04823767
Title: Single Anastomosis Sleeve Iejenal Bypass With Crural Repair in Obese Patient With Hiatus Hernia
Brief Title: Single Anastomosis Sleeve Iejenal Bypass in Obese Patient With Hiatus Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Proffessor, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fac,med 20.3
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single anastomosis sleeve jejunal bypass with hiatal repair (Experimental): Single anastomosis sleeve jejunal bypass with hiatal repair
  Interventions: Other: Single anastomosis sleeve jejunal bypass with hiatal repair

INTERVENTIONS:
Other: Single anastomosis sleeve jejunal bypass with hiatal repair — Single anastomosis sleeve jejunal bypass with hiatal repair

SUMMARY:
single anastomosis sleeve jejunal bypass with hiatal repair for morbid obesity with reflux manifestations

DETAILED DESCRIPTION:
preoperative endoscopy was done and if hiatus hernia was present the patient is undergo single anastomosis sleeve jejunal bypass with hiatal repair for morbid obesity with reflux manifestations

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases
* revisional bariatric procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
the effect of sleeve jejunal bypass on reflux manifestations | 2 months
  evaluation of the effect of sleeve jejunal bypass on reflux manifestations

SECONDARY OUTCOMES:
EWL | one year
  excess weight loss at one year
treatment of comorbidities | one year
  effect on obesity comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Minya, Egypt